CLINICAL TRIAL: NCT07315347
Title: Home Treatment of Patients With Active Cancer and Acute Pulmonary Embolism Without HESTIA Criteria. A Randomised Trial
Acronym: HOME-PEK
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: APHP241014; PHRC-K24-139 (Other Grant/Funding Number: French Ministry of Health); 2025-A01173-46 (Other: ID-RCB)
Record Dates: First submitted 2025-12-18; First posted 2026-01-02 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Active Cancer and Symptomatic or Incidental Pulmonary Embolism Without HESTIA Criteria
Keywords: Active cancer; pulmonary embolism; negative HESTIA rule; home treatment
MeSH Terms: conditions — Pulmonary Embolism

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Home-treatment group (Experimental): Patients will be discharged home within 24hrs after randomisation.
  Interventions: Other: Home-treatment group
- Hospitalisation group (No Intervention): Patients will be admitted in the hospital during at least 48hrs after randomisation. After this time, physicians in charge of the patients will be free to discharge the patients.

INTERVENTIONS:
Other: Home-treatment group — Patients randomised to the home-treatment group will be discharged home within 24hrs after randomisation. Patients will be contacted by the local thrombosis team by phone within 7 days following inclusion.
  Arms: Home-treatment group

SUMMARY:
Main objective of this multisite randomised study aims to demonstrate in patients with active cancer and symptomatic or incidental PE without HESTIA criteria, that home treatment is non-inferior to hospitalisation as regards the 14-day rate of the composite primary endpoint.

Primary endpoint corresponds to the rate of the composite of centrally adjudicated recurrent incidental or symptomatic VTE (i.e. non fatal or fatal PE, proximal and/or distal deep venous thrombosis (DVT) of lower limb or upper limb or catheter-related thrombosis), major or clinically relevant non-major bleeding and all-cause death within 14 days following randomisation. This composite endpoint represents the net clinical benefit of outpatient care.

Included patients will be randomised into two groups and stratified according to symptomatic or incidental PE, site of cancer, localised or metastatic cancer and centre.

Patients randomised to the home-treatment group will be discharged home within 24hrs after randomisation. Patients will be contacted by the local thrombosis team by phone within 7 days following inclusion.

Patients randomised to the hospitalisation group will be admitted in the hospital during at least 48hrs after randomisation. After this time, physicians in charge of the patients will be free to discharge the patients.

DETAILED DESCRIPTION:
Several studies have demonstrated that patients with low-risk pulmonary embolism (PE), selected on simplified PE Severity Index (sPESI) = 0 or without HESTIA criteria, can be safely treated at home. The HOME-PE study demonstrated that HESTIA rule was at least as safe as sPESI score for triaging patients with PE. With both strategies, almost 35% of patients could be managed at home with a low rate of complications (" 1% at Day-30).

PE is a common complication in patients with cancer who are at higher risk for recurrence of venous thromboembolism (VTE), bleeding and PE-related death than patients without cancer. For these reasons, some decision-making tools categorise all patients with cancer at risk of complications and are therefore not eligible for home treatment. In a post hoc analysis of the HOME-PE trial, the 30-day rate of adverse events was higher in patients with active cancer treated at home (4.3%) than in those without (1.0%), but was comparable in patients with cancer hospitalised only because of cancer (3.0%). Home treatment was not a risk factor of complications among cancer patients. Interestingly, 90% of these complications occurred after day-10 suggesting that hospitalisation did not avoid the occurrence of adverse events. Moreover, approximately 50% of PE in patients with cancer is now incidentally detected on imaging undertaken for cancer staging or evaluation of treatment response with a prevalence up to 5%. These patients should be managed in the same manner as symptomatic PE since they have similar prognosis. However, hospitalisation is sometimes challenging in daily practice (availability of bed…) and some of these patients are currently treated at home despite the absence of evidence on the safety of such management.

Home treatment is important for retaining autonomy of patients and may improve their perception of health and quality of life which are particularly relevant for cancer patients. However, this expected benefit have never been confirmed in a prospective trial.

We propose to assess in a randomised controlled trial whether home treatment of patients with active cancer and symptomatic or incidental PE with a negative HESTIA rule is at least as safe as hospitalisation. Furthermore, we will assess the impact of home treatment on several patient-centred outcomes as well as medico-economic issues.

The results are expected to help to define the best management strategy and will provide high level of evidence for cancer associated PE patient care in terms of safety, efficacy and efficiency.

Included patients will be randomised into two groups (1:1) and stratified according to symptomatic or incidental PE, site of cancer, localised or metastatic cancer and centre.

Patients randomised to the home-treatment group will be discharged home within 24hrs after randomisation. Patients will be contacted by the local thrombosis team by phone within 7 days following inclusion.

Patients randomised to the hospitalisation group will be admitted in the hospital during at least 48hrs after randomisation. After this time, physicians in charge of the patients will be free to discharge the patients.

Data will be recorded in a computerised case report form (e-CRF) enabling randomisation between home treatment and hospitalisation. In both groups, physicians in charge of the patients will prescribe anticoagulant according to local protocols. Anticoagulant treatment will be started at the latest immediately after PE diagnosis. All patients will be instructed to contact the local thrombosis team or to report to the ED in case of any new symptoms suggestive of VTE or any bleeding episodes occur. Follow-up will occur at 7, 14, 30 and 90 days after inclusion in both groups to gather clinical events (recurrent VTE, major or clinically relevant bleeding, death), patients-centred outcomes (EQ-5D-5L, PEmbQoL, ACTS) and patients resource utilisation. An independent adjudication committee will evaluate all clinical endpoints blinded to the group allocated.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Symptomatic or incidental hemodynamically stable PE objectively confirmed ≤ 24h according to the ESC guidelines
* Active cancer other than basal-cell or squamous-cell carcinoma of the skin defined at least by one of the followings:
* cancer that has been diagnosed within the past 6 months,
* cancer for which anti-cancer treatment is being given at the time of enrolment or during 6 months before randomisation, or recurrent locally advanced or metastatic cancer
* No HESTIA criteria (i.e. no other medical condition than cancer since cancer is one of the medical condition that can check "yes" to the item).
* For woman of childbearing potential: negative beta-HCG before inclusion
* Signed informed consent
* Affiliated to French " sécurité sociale "
* Good understanding of the French language

Exclusion Criteria:

* Diagnosis of PE established for over 24h before inclusion
* Shock or hypotension defined as systolic blood pressure <90 mmHg or a systolic pressure drop by ≥40 mmHg, for >15 minutes, if not caused by new-onset arrhythmia, hypovolaemia, or sepsis
* Hospitalisation for over 24h
* ECOG performans status 3 or 4
* Impossibility for 30-day follow-up,
* Estimated life expectancy less than 30 days
* Patient in detention by judicial or administrative decision,
* Patient placed under a legal protection measure,
* Patient unable of giving free and informed consent
* Inclusion in another interventional study requiring hospitalisation
* Pregnant or breastfeeding women
* Patient on AME (state medical aid)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 824 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2029-01 (Estimated); Study Completion 2029-03 (Estimated)

PRIMARY OUTCOMES:
Rate of composite primary endpoint | Within 14 days following randomisation
  The rate of the composite of centrally adjudicated recurrent incidental or symptomatic VTE (i.e. non fatal or fatal PE, proximal and/or distal deep venous thrombosis (DVT) of lower limb or upper limb or catheter-related thrombosis), major or clinically relevant non-major bleeding and all-cause death within 14 days following randomisation. This composite endpoint represents the net clinical benefit of outpatient care.
  To assess the non-inferiority of home treatment as compared to hospitalisation, the rates of the composite primary endpoint, at 14 days, will be compared between the two groups using logistic regression adjusted on stratification factors (symptomatic or incidental PE, type of cancer, localised or metastatic cancer, and centre).
  Results will be presented as rates difference (home treatment minus hospitalisation), in this sense.

SECONDARY OUTCOMES:
Key Secondary Endpoint: Change in EQ-5D-5L Index | Inclusion, 7 days, 14 days following randomisation
  Change from baseline in EQ-5D-5L index (5 health dimensions) assessed at inclusion, D7 and D14.
  The EQ-5D-5L system consists of five dimensions (also called items), each exploring one Health-related dimension among mobility, self-care, usual activities, pain/discomfort, anxiety/depression. Each dimension is answered by selecting one of five ordered functional levels (5-levels Likert scale): no problem, slight problems, moderate problems, severe problems, and extreme problems. For each patient, the combination of the five answers corresponds to his/her health state or profile. With the five ordinal levels of each answer encoded 1 to 5 and a total of 3125 possible combinations, "11111" represents full health and "55555" the worst possible health state.
Safety: Rate of Symptomatic or Incidental Recurrent PE and DVT (Lower Limb, Upper Limb, or Catheter-Related) | 7 days, 14 days, 30 days, 90 days following randomisation
  The rate of symptomatic or incidental recurrent PE or proximal and/or distal DVT of lower limb or upper limb or catheter-related.
Safety: Rate of Major Bleeding | 7 days, 14 days, 30 days, 90 days following randomisation
  The rate of major bleeding (ISTH definition).
Safety: Rate of Clinically Relevant Non-Major Bleeding | 7 days, 14 days, 30 days, 90 days following randomisation
  The rate of clinically relevant non-major bleeding.
Safety: Rate of All-Cause Mortality | 7 days, 14 days, 30 days, 90 days following randomisation
  The rate of all-cause mortality.
Safety: Rate of PE-Related Death | 7 days, 14 days, 30 days, 90 days following randomisation
  The rate of PE-related death.
Safety: Rate of Cancer-Related Death | 7 days, 14 days, 30 days, 90 days following randomisation
  The rate of cancer-related death.
Safety: Rate of Patients Meeting EARTH Criteria | 7 days, 14 days following randomisation
  The rate of patients meeting the EARTH criteria, composed by: confirmed new onset of hypoxemia (<90%) requiring oxygen or ventilation support; confirmed new onset of severe hypotension or shock requiring treatment; new confirmed symptomatic cardiac rhythm disorder requiring urgent treatment; symptomatic PE recurrence or symptomatic proximal DVT requiring specific treatment or anticoagulation modification; major bleeding; death possibly related to PE (including death with an unknown cause).
Quality of Life: EQ-5D-5L and EQ VAS | 7 days, 14 days, 30 days, 90 days following randomisation
  The EQ-5D-5L system consists of five dimensions, each exploring one Health-related dimension among mobility, self-care, usual activities, pain/discomfort, anxiety/depression. Each dimension is answered by selecting one of five ordered functional levels (5-levels Likert scale): no problem, slight problems, moderate problems, severe problems, and extreme problems. For each patient, the combination of the five answers corresponds to his/her health state or profile. It also includes a Visual Analogue Scale (VAS) where patients rate their overall health from 0 (worst) to 100 (best).
Quality of Life: PEmbQoL | 30 days, 90 days following randomisation
  Patient-reported Pulmonary Embolism Quality of Life (PEmbQoL) PEmbQoL ordinal scores SL (social limitations), Q2, Q3 and PEmbQoL quantitative scores FO (frequency of Complaints), WR (Work related problems), EC (Emotional complaints), ADL (Activity daily limitation), IO (Intensity of Complaints)
Treatment Satisfaction: Anti-Clot Treatment Scale | 30 days, 90 days following randomisation
  Satisfaction measured using the Anti-Clot Treatment Scale Questionnaire. The Anti-Clot Treatment Scale (ACTS) is a 15-item patient-reported instrument of satisfaction with anticoagulant treatment. It includes a 12-item ACTS Burdens scale and a 3-item ACTS Benefits scale.
Healthcare Resource Utilisation | 14 days, 30 days, 90 days following randomisation
  Mean cumulative hospital length of stay for initial hospitalisation and proportion of patients with unscheduled medical consultations.
Medico-Economic: Cost-Utility and Cost-Effectiveness | 30 days, 90 days following randomisation
  Cost-effectiveness within 30 days and 90 days following randomisation.

CONTACTS AND LOCATIONS:
Overall Officials: Olivier SANCHEZ, MD, Study Chair — Assistance Publique - Hôpitaux de Paris
Locations (20):
- France (20):
  - C12 - Médecine Vasculaire - CHU Amiens Picardie, Amiens
  - C10 - Département médecine urgence - CHU Angers, Angers
  - C08 - Département de Médecine interne et pneumologie - CHU la Cavale Blanche, Brest
  - C11 - Pneumologie - CH René Dubos, Cergy-Pontoise
  - C16 - Département Urgences - CHU Clermont Ferrand, Clermont-Ferrand
  - C05 - Médecine Interne - Hôpital Louis Mourier - APHP, Colombes
  - C13 - Médecine Vasculaire - CHU Dijon, Dijon
  - C04 - Oncologie Médicale - Centre Georges-François Leclerc - CLCC, Dijon
  - C18 - Pneumologie - CH de Versailles Hôpital André Mignot, Le Chesnay
  - C17 - Médecine Interne - CHU Nantes, Nantes
  - C06 - Pneumologie - Hôpital Cochin - APHP, Paris
  - C07 - Médecine Vasculaire - Hôpital Saint Joseph, Paris
  - C01 - Pneumologie et Soins Intensifs - HEGP, Paris
  - C03 - Médecine interne et médecine vasculaire - Hospices Civils de Lyon, Pierre-Bénite
  - C15 - Médecine Interne - CHU Rouen, Rouen
  - C09 - Médecine vasculaire et thérapeuthique - CHU Saint Etienne, Saint-Priest-en-Jarez
  - C19 - Pneumologie - Hôpital Foch, Suresnes
  - C14 - Médecine Vasculaire - CH Toulon, Toulon
  - C20 - Médecine Vasculaire - CHU Toulouse, Toulouse
  - C02 - Département interdisciplinaire d'organisation des parcours patients - Institut gustave Roussy, Villejuif

IPD SHARING:
Plan to Share IPD: Yes
The deindentified individual participant data (IPD) that support the results reported in publications may be shared. Additionally, the IPD outlined in the protocol for a planned meta-analysis may also be made available. A data dictionary defining each field will be made available concurrently with the data transmission.
Supporting Information: Study Protocol, ICF
Time Frame: Two years after the last publication
Access Criteria: Data sharing requires approval from both the sponsor and the principal Investigator (PI), contingent upon a scientific project and the PI team's scientific contribution. The founder may also participate in the decision-making process.
  Teams seeking to acquire IPD must engage with the sponsor and the IP team to discuss the scientific (and commercial) objectives, the specific IP required, the preferred data transmission format, and the proposed timeline. The necessity to inform patients about data sharing or the obligation to undertake procedures with data protection authorities will be evaluated.
  The provision of data through the secure institutional tools of the sponsor AP-HP will be prioritized.
  Technical feasability and financial support considerations will precede the obligatory formalization of a contract, including detailed description of data processing and general and specific security measures.
  The processing must adhere to the European General Data Portection Regulation